CLINICAL TRIAL: NCT06764290
Title: Neural Mechanism Changes in Stroke Patients During Challenging Environments
Brief Title: Neural Changes in Stroke Patients During Challenging Walking Tasks.
Status: Recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhao Jing, Junior physiotherapist, Nanjing Medical University
Other Study IDs: 2024018-1
Record Dates: First submitted 2024-04-10; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: Electroencephalography; gait rehablitation; challenging task
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke participants: Stroke participants with residual abnormal gait.
  Interventions: Other: pedal walking; Other: visual occlusion

INTERVENTIONS:
Other: pedal walking — Pedal walking is a challenging walking task that can be used as a form of physical therapy for stroke participants.
Other: visual occlusion — Walking with eyes-covered is a challenging walking task that can be used as a form of physical therapy for stroke participants.

SUMMARY:
For stroke patients, a challenging, unfamiliar, and more difficult task may increase the likelihood of brain activation to stimulate recovery. Pedal walking and walking with eyes-covered are both difficult and challenging tasks for stroke patients. The investigators intend to study the biomechanics and neural mechanisms of challenging pedal walking and walking with eyes covered.

Stroke participants will wear electroencephalogram electrode caps and perform three tasks: walking on a flat surface for 60 seconds, walking on pedal for 60 seconds, and walking with eyes covered for 60 seconds.

DETAILED DESCRIPTION:
Stroke participants will wear a 32-lead electroencephalogram electrode cap (Zhentai Technology Company, Xi 'an, China), first walk on a flat ground for 60 seconds, rest for 2 minutes, then walk on the pedal for 60 seconds, rest again for 2 minutes, and walk for 60 seconds with eyes-covered.

ELIGIBILITY:
Inclusion Criteria:

* First-time occurrence of stroke confirmed by computed tomography or magnetic resonance imagingClinical diagnosis of stroke
* Disease duration of more than 14 days， less than 1 year
* Able to walk independently but with a lingering abnormal gait

Exclusion Criteria:

* Lesions accumulate in the brainstem
* Lesions accumulate in the cerebellum
* Impaired vision
* Severe cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients, including outpatients and inpatients.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Weight Phase Lag Index | The study was an observational cross-sectional study with data collected at the same time as the trial was being conducted, so the duration was 60 seconds
  The Weighted Phase Lag Index (WPLI) is a measure used to quantify phase synchronization in electrophysiological data.Continuously measure the connectivity of the coupling of neural oscillatory activity in the brain, while being statistically more powerful in detecting changes in signal phase synchronization.The WPLI ranges from 0 to 1, with 0 indicating no phase synchronization and 1 indicating complete phase synchronization.
Relative power | The study was an observational cross-sectional study with data collected at the same time as the trial was being conducted, so the duration was 60 seconds
  The electroencephalogram signal in the time domain is converted into the relevant information in the frequency domain, the frequency bands are divided, and the relative power results of each channel in each frequency band are derived. Among them, delta:1-4Hz, theta:4-8Hz, alpha:8-15Hz, beta:15-30Hz, gamma:30-45Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li Zhang, doctor, Study Director — Geriatric Hospital of Nanjing Medical University
Locations (2):
- China (2):
  - Geriatric Hospital of Nanjing Medical University, 269 Qingmen Street, Nanjing, Jiangsu
  - Geriatric Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after publication.
Access Criteria: Request from the corresponding author by email.

REFERENCES:
- [Background] Krakauer JW. Motor learning: its relevance to stroke recovery and neurorehabilitation. Curr Opin Neurol. 2006 Feb;19(1):84-90. doi: 10.1097/01.wco.0000200544.29915.cc. PMID 16415682
- [Background] Fettrow T, Hupfeld K, Tays G, Clark DJ, Reuter-Lorenz PA, Seidler RD. Brain activity during walking in older adults: Implications for compensatory versus dysfunctional accounts. Neurobiol Aging. 2021 Sep;105:349-364. doi: 10.1016/j.neurobiolaging.2021.05.015. Epub 2021 May 31. PMID 34182403
- [Background] Kulkarni A, Cui C, Rietdyk S, Ambike S. Humans prioritize walking efficiency or walking stability based on environmental risk. PLoS One. 2023 Apr 7;18(4):e0284278. doi: 10.1371/journal.pone.0284278. eCollection 2023. PMID 37027387
- See also: This paper suggests that the rehabilitation of stroke patients may require more challenging tasks — http://pubmed.ncbi.nlm.nih.gov/16415682/
- See also: This paper suggests that the performance of complex walking tasks may involve top-down cortical control in the brain centers — http://pubmed.ncbi.nlm.nih.gov/34182403/
- See also: This paper shows that the central nervous system will actively respond to environmental changes and adjust to obtain stable motor output — http://pubmed.ncbi.nlm.nih.gov/37027387/